CLINICAL TRIAL: NCT01107782
Title: Phase 2 Study of Fetal Growth Retardation Treatment by Sildenafil
Brief Title: Sildenafil and Uteroplacental Perfusion
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Marzieh Vahid Dastjerdi, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 87-821
Record Dates: First submitted 2010-01-13; First posted 2010-04-21 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Fetal Growth Retardation
Keywords: sildenafil; FGR
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil (Experimental)
  Interventions: Drug: sildenafil
- Placebo control (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — 50 mg TDS orally until birth
  Other Names: viagra
  Arms: sildenafil
Drug: placebo — 50mg tid
  Other Names: placebo tid
  Arms: Placebo control

SUMMARY:
The purpose of this study is to determine whether sildenafil is effective and safe in the treatment of fetal growth restriction.

DETAILED DESCRIPTION:
Fetal growth retardation affects up to 8% of all pregnancies and has massive short term (increased fetal morbidity and mortality) and long-term (increased incidence of cardiovascular disorders in adulthood) health implications.

Doppler waveform analysis of these pregnancies suggests compromised uteroplacental circulation and placental hypoperfusion.

Our aim is to assess if sildenafil citrate could improve vasodilatation in FGR pregnancies.

Sildenafil citrate may offer a potential therapeutic strategy to improve uteroplacental perfusion in FGR.

Animal studies suggest that phosphodiesterase-5 (PDE5) inhibitors, such as sildenafil citrate, may improve uterine blood flow .

ELIGIBILITY:
Inclusion Criteria:

* FGR pregnancies in 24-37 weeks of GA

Exclusion Criteria:

* vasodilator agents usage
* history of cardiovascular morbidity specially of right heart side
* drug or alcohol abusers
* systolic BP more than 210 mm Hg or diastolic BP more than 120 mm Hg

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Uteroplacental Perfusion | 2 hours after sildenafil ingestion

SECONDARY OUTCOMES:
fetal growth | after 6 months
umbilical artery blood gass assessment | immediately after birth
effect on fetal well being | 2 hours after sildenafil
  when BP score is<8 we repeat it after sildenafil ingestion

CONTACTS AND LOCATIONS:
Overall Officials: marzieh vahid dastjerdi, M.D., Study Chair — Iranian's ministery of health; Sayedeh Afagh Hosseini, MD., Study Director — resident of OB&GYN
Locations (1):
- Tehran UMS, Tehran, Tehran Province, Iran